CLINICAL TRIAL: NCT03385200
Title: Contrast-enhanced Ultrasound in Neoadjuvant Chemotherapy of Breast Cancer
Brief Title: KVUS at Neoadjuvant CTx of Breast Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: RWTH Aachen University (Other)
Collaborators: Univ.-Prof. Dr. med. F. Kiessling (Unknown)
Responsible Party: Principal Investigator, Elmar Stickeler, Univ.-Prof. Dr. med., RWTH Aachen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-134
Record Dates: First submitted 2017-12-19; First posted 2017-12-28 (Actual); Last update posted 2017-12-28 (Actual); Status verified 2017-12

CONDITIONS: Early Primary Breast Cancer
Keywords: breast cancer, neoadjuvant chemotherapy, ultrasound, microbubbles
MeSH Terms: conditions — Breast Neoplasms | interventions — contrast agent BR1

STUDY DESIGN:
Intervention Model Description: Parellel Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- A (Active Comparator): Application and measurement of tumor size using contrast agent-enhanced diagnostic and therapy supporting (with SonoVue®) ultrasound
  Interventions: Drug: SonoVue
- B (No Intervention): Application and measurement of tumor size using contrast agent-enhanced diagnostic ultrasound

INTERVENTIONS:
Drug: SonoVue — As part of the study therapy supportive ultrasound will be performed with iv Infusion of the chemotherapeutic agent.
  Arms: A

SUMMARY:
Effect of the contrast-enhanced diagnostic ultrasound during neoadjuvant chemotherapy of breast cancer on the achieved tumor size reduction and tolerability of chemotherapy

DETAILED DESCRIPTION:
The 5-year survival rate of breast cancer patients is decreasing in the advanced, metastatic stage from 99% to 26%. Therefore an optimization of the therapy of advanced breast cancer is urgently needed.

To increase the echogenicity of the blood in the ultrasound, microbubbles were developed working as stable, biocompatible contrast agent in ultrasound. Such a clinically approved ultrasound contrast agent is SonoVue® (Bracco International B.V., Amsterdam). SonoVue® is approved by the European Medicines Agency (EMA) (approval number EU/1/01/177/002) for the visualization of focal vascularization lesions of the liver and breast within Doppler sonography and is applied in breast cancer patients primarily for the purpose of diagnosis as well as to evaluate the response to the neoadjuvant used chemotherapy.

Animal studies using the contrast enhanced ultrasound have shown that the administration of this contrast agent increases the penetration and accumulation of drugs in the tumor as well as the permeability of the blood-brain barrier resulting in a precise and effective drug distribution. In the tumor animal model it could be shown that a combined treatment with chemotherapy and contrast enhanced ultrasound results in a decreased tumor growth and a prolonged survival. Patients with inoperable pancreatic cancer showed a reduced tumor growth and better tolerability of chemotherapy when administrating the contrast enhanced diagnostic ultrasound during palliative chemotherapy. This could be due to the better tumor response, but also due to the more targeted chemotherapy distribution.

The purpose of this study is to examine whether the use of the contrast enhanced diagnostic ultrasound during neoadjuvant chemotherapy results in an increased tumor regression in comparison to native ultrasound. It is an Investigator Initiated Trial and is funded by internal means.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent
* age > 18 yrs
* histologically confirmed primary breast cancer including all intrinsic subtypes
* treatment with neoadjuvant chemotherapy
* persons who are legally competent and mentally able to follow the instructions of the study team

Exclusion Criteria:

* hypersensitivity / allergy to sulfur hexafluoride, Macrogol 4000, distearoylphosphatidylcholine, dipalmitoylphosphatidylglycerol-sodium, palmitic acid
* right-left shunt,
* severe pulmonary hypertension (pulmonary arterial pressure > 90 mmHg)
* uncontrolled systemic hypertension
* acute respiratory distress syndrome
* pregnancy
* commitment of the patient to any resident institution by order of any court or authority
* expectation of missing compliance
* alcohol or drug abuse
* patients who are in a relationship of dependence or in a working relationship to the sponsor, the investigator or his representative

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-12-12 (Actual); Primary Completion 2019-06-12 (Estimated); Study Completion 2019-12-12 (Estimated)

PRIMARY OUTCOMES:
Tumor size reduction (1) | 18 / 24 weeks
  pCR (pathohistological complete remission)
Tumor size reduction (2) | 18 / 24 weeks
  cCR (clinical complete remission)
Tumor size reduction (3) | 18 / 24 weeks
  measured by ultrasound (% reduction in therapy)

SECONDARY OUTCOMES:
proliferation rate of the tumor cells | 18 / 24 weeks
  Ki67 protein analysis
narrowing the invasion front of the tumors | 18 / 24 weeks
  ultrasound
macrophage density in the tumor | 18 / 24 weeks
  serum chemistry
vascularization of the tumor | 18 / 24 weeks
  ultrasound
tolerability of chemotherapy | 18 / 24 weeks
  % reduction in therapy

CONTACTS AND LOCATIONS:
Overall Officials: Elmar Stickeler, niv.-Prof. Dr. med., Principal Investigator — Department of Gynecology and Obstetrics
Locations (1):
- Department of Gynecology and Obstetrics, Aachen, Germany

IPD SHARING:
Plan to Share IPD: Undecided
The study results will be published in at least one scientific article.